CLINICAL TRIAL: NCT01333137
Title: An Open-Label Randomized Phase II Trial Comparing Gemcitabine and Carboplatin With and Without P276-00 in Subjects With Metastatic Triple Negative Breast Cancer, With a Phase I Run-in of Escalating Dose of P276-00 Added to Gemcitabine and Carboplatin
Brief Title: A Clinical Trial Comparing Gemcitabine and Carboplatin With and Without P276-00 in Subjects With Metastatic Triple Negative Breast Cancer, With a Run-in of Escalating Dose of P276-00 Added to Gemcitabine and Carboplatin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P276-00/52/10
Record Dates: First submitted 2011-04-08; First posted 2011-04-11 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Breast Cancer
Keywords: Triple negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine and Carboplatin (Active Comparator): Gemcitabine 1000 mg/m2/day on Days 1 & 8 and carboplatin at AUC 2 on Days 1 and 8 every 21 days.
  Interventions: Drug: Gemcitabine and Carboplatin
- P276-00 along with Gemcitabine and carboplatin (Experimental): P276-00 will be administered at starting dose of 100 mg/m2/day (and higher if tolerated) in 200 mL of 5% dextrose as an iv infusion over 30 minutes, on Days 1 to 5, along with gemcitabine 1000 mg/m2/day and carboplatin at AUC 2 on Days 1 & 8 every 21 days.In Phase 2 component, P276-00 will be administered at recommended phase II dose of P276-00 in combination with standard dose of gemcitabine and carboplatin.
  Interventions: Drug: P276-00 along with Gemcitabine and carboplatin

INTERVENTIONS:
Drug: Gemcitabine and Carboplatin — Gemcitabine 1000 mg/m2/day on Days 1 & 8 and carboplatin at AUC 2 on Days 1 and 8 every 21 days.
  Arms: Gemcitabine and Carboplatin
Drug: P276-00 along with Gemcitabine and carboplatin — In phase I run in period, P276 00 will be administered at starting dose of 100 mg/m2/day (and higher if tolerated) in 200 mL of 5% dextrose as an iv infusion over 30 minutes, on Days 1 to 5, along with gemcitabine 1000 mg/m2/day and carboplatin at AUC 2 on Days 1 & 8 every 21 days. In Phase 2 component, P276-00 will be administered at recommended phase II dose of P276-00 in combination with standard dose of gemcitabine and carboplatin.
  Arms: P276-00 along with Gemcitabine and carboplatin

SUMMARY:
P276-00 is a novel, potent, small-molecule, flavone-derived Cdk 4 D1, Cdk1 B, and Cdk9 T inhibitor, with potent cytotoxic effects against chemosensitive and chemoresistant cancer cell lines.This study is planned to compare efficacy of the standard chemotherapy regimen of gemcitabine and carboplatin when administered with or without P276-00 in subjects with advanced triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Females of age ≥18 years.
2. Histologically documented metastatic triple negative breast cancer (any triple negative breast cancer for Phase I)
3. Two or fewer chemotherapy regimens for advanced disease (no limit of prior regimens for Phase I)
4. ECOG performance score of 1 or less
5. Presence of measurable disease by RECIST 1.1 criteria (not for the Phase I portion)
6. Ability to understand and the willingness to sign a written informed consent document (ICD)
7. Full recovery from all prior treatment toxicities to Common Terminology Criteria for Adverse Events (CTCAE V.4) Grade ≤ 1

Exclusion Criteria:

1. Prior chemotherapy or biologic/targeted anticancer agents within 4 weeks of study drug administration
2. Prior radiation therapy within 6 weeks of study drug administration
3. Subject with known active CNS metastases and/or carcinomatous meningitis. However, subjects with CNS metastases who have completed a course of therapy would be eligible for the study provided they are clinically stable for at least 1 month prior to entry as defined as: (1) no evidence of new or enlarging CNS metastasis or new neurological symptoms attributable to CNS metastases (2) off steroids that are used to minimize surrounding brain edema.
4. Prior therapy with gemcitabine or a platinum agent (not for the Phase I part)
5. Prior therapy with a Cdk/cyclin inhibitor or any flavones derivative
6. QTc interval >450 msec (using Fridericia's formula)
7. Any acute illness including uncontrolled diabetes, symptomatic or otherwise uncontrolled cardiac disease (coronary artery disease, arrhythmias, congestive heart failure) or other illness that in the judgment of the investigator would introduce additional medical risks
8. Visceral crisis including extensive liver disease with>50% parenchymal involvement or lymphangitic pulmonary disease
9. History of other prior malignancies except for properly treated basal cell or squamous cell carcinoma of skin, in situ cervical cancer, or in situ breast cancer
10. Expected survival of less than 3 months
11. Hemoglobin <9.0 gm/dL
12. Absolute neutrophil count <1500/mm3
13. Platelet count <100,000/mm3
14. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >3 × institutional upper limit of normal (ULN)
15. Total bilirubin, >1.5 × institutional ULN
16. Serum creatinine >1.5 mg/dL
17. Subjects with known infection with human immunodeficiency virus (HIV), tuberculosis, Hepatitis C or Hepatitis B
18. Pregnant or lactating women
19. Women of childbearing potential not willing to use approved methods of contraception after signing the ICD, during the entire study and for at least 4 weeks after completion of study or following withdrawal from the study

    -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Median Progression free survival | 1 year and above
  The primary efficacy endpoint will be median progression-free survival (PFS), defined as the time from the beginning of study treatment to the occurrence of documented disease progression or recurrence, or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | at 3 years
Overall survival at 6 months | at 6 months
Progression Free Survival at 6 months | at 6 months
Objective response rate | upto 3 years and above
Duration of response | upto 3 years and above

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Debasish Tripathy, Principal Investigator — USC/Norris Comprehensive Cancer Center 1441 Eastlake Avenue, Rm 3440, Los Angeles, CA 90033
Locations (4):
- United States (4):
  - Disney Cancer Center, Burbank, California
  - 3855 Health Sciences Drive, La Jolla, California
  - UC Davis Cancer Center, Sacramento, California
  - Washington University, St Louis, Missouri